CLINICAL TRIAL: NCT02422108
Title: Denosumab and Male Infertility: a Prospective Intervention Study
Brief Title: TNFSF11 Inhibition and Fertility: a Prospective Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Martin Blomberg Jensen (Other)
Responsible Party: Sponsor-Investigator, Martin Blomberg Jensen, Senior Researcher, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBG-study2; H-15001992 (Other: The Regional Committee on Biomedical Research Ethics)
Record Dates: First submitted 2015-04-06; First posted 2015-04-21 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Testis; Infertility; Sperm
Keywords: RANKL
MeSH Terms: conditions — Infertility | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intervention (Experimental): Denosumab (Prolia) 60 mg s.c.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab
  Other Names: Prolia

SUMMARY:
The receptor activator of NF-kB ligand (RANKL) system is considered important for bone homeostasis and comprises three important factors. RANKL exist in three isoforms but the predominant function is mediated by the transmembrane ligand that binds to a specific receptor (receptor activator of NF-KB (RANK)) on a neighbour cell that subsequently activates NFKB and regulates cell cycle OPG is an endogenous secreted protein that binds RANKL and inhibits its signalling.

Thus, the RANK/RANKL system is vital for activation of the bone resorbing cells (osteoclasts). In bone the bone synthesizing cells (osteoblasts) express RANKL that signals to RANK on the immature osteoclasts. This induces proliferation and activation of the cells they start to proliferate and resorp bone. OPG is produced by somatic cells in the bone and this production is regulated by sex hormones, TGF-B and various other substances. Today a human made recombinant antibody against RANKL, Denosumab is used to treat osteoporosis as it inhibits RANKL signalling and thus causes less bone resorption in humans.

RANKL, RANK and OPG are expressed in the testis and this pathway appears to be a novel regulator of germ cell proliferation. Decreased semen quality is a major factor of male infertility. Semen quality is a measure of the ability of the sperm to accomplish fertilization. Evaluation of male fertility potential is today basically conducted through semen analysis. There is no treatment for men with no sperm in the ejaculate and there exist no drug that can increase sperm counts.Therefore, drugs that can lower RANKL expression/activity for instance an antibody against RANKL such as Denosumab may be used for this new indication: A new treatment option of infertile men with impaired semen quality.

DETAILED DESCRIPTION:
The receptor activator of NF-kB ligand (RANKL) system is considered important for bone homeostasis . RANKL exist in three isoforms and the effects of all isoforms are mediated through binding to a specific receptor (receptor activator of NF-KB (RANK)). RANKL is predominantly found as a transmembrane protein and signalling is therefore dependent on cell-cell interaction to a neighbouring cell expressing RANK that subsequently activates NFKB and regulates cellular activation through regulation of cell cycle i.e proliferation, differentiation and apoptosis. RANKL-RANK interaction is modified by osteoprotegerin (OPG), which is an endogenous secreted protein that binds RANKL and inhibits its signalling.

RANK/RANKL triggers a network of TRAF-mediated kinase cascades that promote osteoclast differentiation. RANKL is expressed on osteoblast cells and its receptor, Rank, on pre- osteoclastic cells. RANKL expression is stimulated by a number of factors, such as IL-1 , IL-6, IL-11 , IL-17, TNF- α, vitamin D, Ca2+, parathyroid, glucocorticoids, prostaglandin E2, and immunosuppressive drugs, and is down-regulated by TGF-α. The RANK/RANKL interaction induces differentiation and formation of multinucleated mature osteoclasts, causing bone resorption. The third protein agonist, osteoprotegerin (OPG), is also produced by osteoblasts and is known to exert an inhibitory effect on the pre-osteoclastic differentiation process. By binding to RANKL also known as osteoprotegerin binding protein (OPGbp), OPG inhibits the RANK/RANKL interaction and subsequent osteoclastogenesis. OPG is thus a very efficient anti-resorptive agent. It also serves as a decoy receptor for the tumour necrosis factor-related apoptosis-inducing ligand (TRAIL) and increases cell survival by blocking the apoptotic effects of this ligand. The fact that the overexpression of OPG in mice results in severe osteopetrosis and that OPG-null mice are osteoporotic is testimony to the physiological importance of OPG. The lack of RANK or RANKL induces osteopetrosis in mice.

Thus, the RANK/RANKL system is vital for activation of the bone resorping cells (osteoclasts). In the skeleton the bone synthesizing cells (osteoblasts) express RANKL that signals to RANK on the immature osteoclasts. This induces proliferation and activation of the cells they start to proliferate and resorp bone. OPG is produced by somatic cells in the bone and this production is regulated by sex hormones, TGF-B and various other substances. Today a human made recombinant antibody against RANKL, Denosumab is used to treat osteoporosis as it inhibits RANKL signalling and causes less bone resorption in humans. RANKL signalling has only two other known additional functions in healthy humans where it is involved in lactation and the immune response.

The investigators have data showing that RANKL, RANK and OPG are expressed at both RNA and protein level in the human testis. The Sertoli cells express RANKL, while the germ cells express RANK and the peritubular cells express OPG. Normally, RANKL activates NFKB and activation of this pathway in the male gonad appears to regulate whether the testicular cells proliferate or undergo apoptosis in the testis. The investigators' in vitro, ex vivo and in vivo data from functional models support this suggestion and this pathway appears therefore to be a novel regulator of germ cell proliferation.

Decreased semen quality is a major factor of male infertility. Semen quality is an indirect measure of the ability of the sperm to accomplish fertilization. Evaluation of male fertility potential is evaluated by semen analysis. Semen analysis evaluates certain characteristics and the most common variables measured to evaluate sperm quality are: sperm count, motility and morphology.

There is no treatment for men with no spermatozoa in the ejaculate or even a drug that can increase sperm number in infertile men.Therefore, we suggest that antibodies against RANKL such as Denosumab, may be used as a novel treatment option for male infertility , which highlights a new indication for Denosumab treatment.

The investigators will therefore test whether inhibition of RANKL by Denosumab in humans increases sperm production and semen quality in this small prospective intervention study.

We will invite 15 infertile men for detailed screening to secure inclusion and study completion of anticipated 12 infertile men

BIOSTATISTICAL ANALYSIS

All the analyses will be performed according to Good Clinical Practice guidelines and the primary analyses in the intention-to-treat population, which included all patients who received the first dose of medicine on day 1. We will analyze the data in two ways. The primary analysis will proceed according to baseline values compared with outcomes variables after intervention. The secondary analysis will be based on stratifying the men according to subgroup analyses in relation to the predefined primary and secondary endpoints.

Data analysis and quality The primary end points for this protocol will be changes in sperm production evaluated by total sperm number, sperm concentration followed by number of progressive and motile sperm, morphologically normal sperm, sperm motility, progressive motility and morfology which will be compared by paired t-test. Multiple secondary endpoints exist but for the initial investigation focus will be on changes of the following secondary endpoints: Sperm DFI, FSH, Inhibin B, serum OPG, RANKL, OPG, vitamin D and calcium homeostasis. Subjects who terminate participation after visit day 1 but before visit day 180 will be included for data analysis up to the last day they provided semen and bloodsample. Men that only deliver semen samples occasionally or have missing data at any visit will still be included in the analysis. Men that do not meet the criteria in the protocol will be excluded from the analysis. Men with fever above 38.5 degrees Celsius will not be included in the analyses up to 3 months after the fever episode. Semen samples obtained with an abstinence period less than 24 hours or with a semen volume < 1.5 ml will not be included in the analyses. Those values will then be carried forward for analyses. A significance level of 5% is used. For the primary analyses Bonferronu-Holm p-value correction is calculated additionally. For the secondary analysis no multiple test correction are used. Instead results are discussed in view of the multiple testing situations.

1. Analyses between baseline versus different timepoints The first step will be to compare the changes in primary outcomes between baseline versus the different timepoints. Spermatogenesis normally takes up to 70 days in men and we will therefore determine the difference to all the individual timepoints and calculate average for days 80, 120 and 180 and compare with baseline values to determine the effect of RANKL inhibition on the whole length of spermatogenesis. This analysis will show if there is a significant difference between groups. For outcomes measured repeatedly, this will entail comparing the estimated slopes, or rates of change, of each outcome between the groups. Mixed models allow for the correlation between the repeated observations baseline-day 1-day 80- day 180 from each man to be suitably incorporated into parameter estimation. For all endpoints measured at baseline and day 180, paired t-tests will be used to assess there is a significant difference between the groups and determine whether the mean change within each group differs significantly from zero. In both cases, data will be transformed as necessary to meet model assumptions. Afterwards, the same analysis will be conducted by using multiple regression with relevant confounders such as season, BMI, smoking, duration of abstinence, time from ejaculation to motility assessment, fever etc. to see if this changes the results For outcomes measured that cannot be compared with t-test or other parametric tests at day 1, day 80 and day 180, groups will be compared using non-parametric tests such as Wilcoxon Mann-Whitney test. For Binary outcome the data will be compared between the two groups by means of conditional logistic-regression analysis with adjustment for relevant confounders (defined as being significantly p<0.05 associated).
2. Analyses after stratification into subgroups Subjects will be grouped according to their BMI, semen quality, serum RANKL, OPG, calcium, PTH, osteocalcin or other bonefactors evaluated at the day of screening. The subgroup analyses will in accordance with normal clinical practice and stratification in appropriate groups according to the clinical (BMI <25, 25-30, >30 etc.), tertiles or highest/lowest versus remaining at baseline. Analyses will be performed on each timpeoint compared with baseline in addition to mean/median of visit day 80, 120, 180 with baseline and mean/median of all visits after intervention.

ELIGIBILITY:
Infertile men referred for evaluation of male infertility at department of growth and reproduction or infertile men interested in participation in clinical trials.

Inclusion Criteria:

* Male with an age > 18 years old
* Referred for male infertility with sperm concentration >= 0.1 million/ml.
* Additionally, all men must have either sperm concentration < 20 million/ml or < 50% progressive motile spermatozoa or < 12% morphological normal spermatozoa using strict criteria

Exclusion Criteria:

Men with chronic diseases such as

* diabetes mellitus
* Thyroid disease
* endocrine disturbances in need of treatment
* malignant disease
* or diseases known to interfere with calcium homeostasis (such as inflammatory disease with granuloma: sarcoidoses, tuberculosis, Wegeners, vasculitis, inflammatory bowel disease (Crohn's and colitis ulcerosa etc).
* Men with previous testis cancer
* If there is an indication for testis biopsy and it is planned or conducted within the next 6 months
* Serum 25-hydroxy-D3 < 50 nmol/l
* Serum Calcium ion < 1,18 or > 1,35 mmol/l
* Serum OPG >4 pg/ml
* Serum PTH <1.6 or >6 pmol/l
* Inhibin-B < 50 pg/ml
* Latex Allergy
* no good oral condition or major implants
* BMD < -1,5 in columna lumbalis and collum femoris

Criteria for drop out:

* Abrogation of the treatment
* Newly diagnosed endocrine, calcium metabolic disease, parathyroid, thyroid, diabetes or other endocrine disease in need of treatment
* New malignant disease
* Treatment with chemotherapy, immunomodulating therapy, salazopyrin
* Oral or iv treatment with steroid hormones
* New treatment with diuretics, antihypertensive treatment, treatment the heart, calcium channel blockers
* If testis biopsy is performed or other surgery in the genital region during the trial
* Prolia Intoxication

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05; Primary Completion 2017-02 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in sperm production | after 5, 20, 40, 80, 120, 180 days
  evaluated by determining total sperm count and sperm concentration

SECONDARY OUTCOMES:
change in sperm DNA fragmentation index | after 20 and 120 days
  DNA fragmentation
change in number of motile sperm | after 5, 20, 40, 80, 120, 180 days
  multiplying the percentage of motile sperm with total sperm count and similar for progressive motile sperm
change in number of morphological normal sperm | after 5, 20, 40, 80, 120, 180 days
  multiplying the percentage of morphological normal sperm with total sperm count
change in sperm motility | after 5, 20, 40, 80, 120, 180 days
  motilility (ABC) and progressive motility (AB)
change in semen morphology | after 5, 20, 40, 80, 120, 180 days
  morphology
change in semen volume | after 5, 20, 40, 80, 120, 180 days
  volume
change in Inhibin B | after 5, 20, 40, 80, 120, 180 days
  Change in inhibin B, Inhibin B/FSH ratio
change in sex hormones or gonadotropins | after 5, 20, 40, 80, 120, 180 days
  testosterone, estradiol, INSL3, AMH, progesterone, LH, FSH
change in BMD | after180 days
  lumbar spine and collum femoris
Change in vitamin d metabolites | after 5, 20, 40, 80, 120, 180 days
  25-OHD, 1,25OHD, 24,25OHD,
change in seminal plasma concentrations of RANKL, OPG, RANK | after 5, 20, 40, 80, 120, 180 days
change i serum PTH, alkaline phosphatase, calcium, phosphate, | after 5, 20, 40, 80, 120, 180 days
change i serum FGF23, Klotho, osteocalcin, osteopontin, calcitonin, pnp, procollagen III, OPG, RANKL, Sclerostin and other bone markers | after 5, 20, 40, 80, 120, 180 days
change in the number of spermatozoa expressing CYP24A1, VDR or RANKL | after 5, 20, 40, 80, 120, 180 days
change in seminal plasma levels of pH,HCO3, calcium, zink, phosphat, FGF23, Klotho, osteocalcin, osteopontin. | after 5, 20, 40, 80, 120, 180 days
change in seminal plasma levels of FGF23, Klotho, osteocalcin, osteopontin. | after 5, 20, 40, 80, 120, 180 days
change in bloodpressure. | after 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Martin M Blomberg Jensen, MD, DMSc, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Anastasilakis AD, Toulis KA, Goulis DG, Polyzos SA, Delaroudis S, Giomisi A, Terpos E. Efficacy and safety of denosumab in postmenopausal women with osteopenia or osteoporosis: a systematic review and a meta-analysis. Horm Metab Res. 2009 Oct;41(10):721-9. doi: 10.1055/s-0029-1224109. Epub 2009 Jun 17. PMID 19536731
- [Background] Anastasilakis, A. D., et al.
- [Background] Anastasilakis AD, Toulis KA, Polyzos SA, Terpos E. RANKL inhibition for the management of patients with benign metabolic bone disorders. Expert Opin Investig Drugs. 2009 Aug;18(8):1085-102. doi: 10.1517/13543780903048929. PMID 19558335
- [Background] Blomberg, Jensen M.
- [Background] one, H. G., et al.
- [Background] Boonen, S., et al.
- [Background] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655
- [Background] Jorgensen, A., et al.
- [Background] Kwiecinski GG, Petrie GI, DeLuca HF. Vitamin D is necessary for reproductive functions of the male rat. J Nutr. 1989 May;119(5):741-4. doi: 10.1093/jn/119.5.741. PMID 2723823
- [Background] Papapoulos, S., et al.
- [Background] Polyzos, S. A., et al.
- [Background] Schwarz, P., et al.
- [Background] Skakkebaek NE, Rajpert-De Meyts E, Main KM. Testicular dysgenesis syndrome: an increasingly common developmental disorder with environmental aspects. Hum Reprod. 2001 May;16(5):972-8. doi: 10.1093/humrep/16.5.972. PMID 11331648
- [Background] Toulis KA, Anastasilakis AD. Increased risk of serious infections in women with osteopenia or osteoporosis treated with denosumab. Osteoporos Int. 2010 Nov;21(11):1963-4. doi: 10.1007/s00198-009-1145-1. Epub 2009 Dec 15. No abstract available. PMID 20012939
- [Background] Uhland AM, Kwiecinski GG, DeLuca HF. Normalization of serum calcium restores fertility in vitamin D-deficient male rats. J Nutr. 1992 Jun;122(6):1338-44. doi: 10.1093/jn/122.6.1338. PMID 1588451